CLINICAL TRIAL: NCT01469871
Title: Reduction of Tape Blisters After Hip Surgery. A Prospective Evaluation of Three Types of Dressings.
Brief Title: Evaluation of Three Types of Dressings After Hip Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Pelet Stephane, Dr Stephane Pelet MD, PhD Orthopedic surgeon, Hopital de l'Enfant-Jesus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEJ-481
Record Dates: First submitted 2011-11-04; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Tape Blisters; Hip Surgery
Keywords: Dressing; Blisters; Silicone
MeSH Terms: conditions — Blister | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hypafix Transparent dressing (Active Comparator): The Hypafix Transparent dressing, a stretchable dressing, will be used to treat the patients in this group
  Interventions: Device: Dressing of wound
- Mepore Pro dressing (Active Comparator): The Mepore Pro dressing, a self-adhesive perforated dressing, will be used to treat the patients in this group
  Interventions: Device: Dressing of wound
- Mepilex Border dressing (Active Comparator): The Mepilex Border dressing, a self-adherent soft silicone dressing, will be used to treat the patients in this group
  Interventions: Device: Dressing of wound

INTERVENTIONS:
Device: Dressing of wound — The wound will be dressed using the Hypafix Transparent dressing after hip surgery.
  Arms: Hypafix Transparent dressing
Device: Dressing of wound — The wound will be dressed using the Mepore Pro dressing after hip surgery.
  Arms: Mepore Pro dressing
Device: Dressing of wound — The wound will be dressed using the Mepilex Border dressing after hip surgery.
  Arms: Mepilex Border dressing

SUMMARY:
The purpose of this study is to determine if one of the new types of dressings (MEPORE PRO and/or MEPILEX BORDER ) will reduce the blister rate compared to the currently used HYPAFIX.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 45 years old or older
* Hip surgery at Hopital de l'Enfant-Jesus between 02/2009 and 01/2010 (THR,rTHR, DHS, screw fixation, hemiarthroplasty, resurfacing)
* Signed consent form

Exclusion Criteria:

* Allergy to dressing
* Polytrauma / high energy trauma
* Wound at the surgical site prior to surgery
* Neurological deficit of operated side (hemiplegia, etc.)
* Bilateral fracture

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of tape blisters after hip fracture surgery | Participants will be followed for the duration of hospital stay, an expected average of 8 days

SECONDARY OUTCOMES:
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 8 days
The correlation between risk factors and tape blisters | Participants will be followed for the duration of hospital stay, an expected average of 8 days
The possible link between the presence of tape blisters and hospital morbidity. | Participants will be followed for the duration of hospital stay, an expected average of 8 days
The costs related to a tape blister. | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  The actual costs related to a tape blister will be calculated by adding the costs of additional dressings, the costs associated with an extended hospital stay and the additional costs associated with the use of external resources.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Pelet, MD,PhD, Principal Investigator — Hopital l'Enfant-Jésus
Locations (1):
- Centre hospitalier affilié universitaire de Quebec - Hopital l'Enfant-Jesus, Québec, Quebec, Canada